CLINICAL TRIAL: NCT06377722
Title: Phase II Study for the Evaluation of Neoadjuvant Treatment With Cabozantinib Pior to Cytoreductive Nephrectomy in Patients With Advanced or Metastatic Renal Cells Cancer
Brief Title: Cabozantinib Treatment Prior to Cytoreductive Nephrectomy in Patients With Advanced or Metastatic Renal Cells Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The achieved number of samples has been smaller than the planned 50 thus, a mainly descriptive final result analysis was conducted, as presented herein.
Sponsor: Fundacion Oncosur (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABOPRE
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Renal Cell Carcinoma Metastatic; Renal Cell Carcinoma Stage IV; Renal Cell Carcinoma Stage III
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with cabozantinib prior to cytoreductive nephrectomy (Experimental): To evaluate the efficacy of preoperative cabozantinib treatment as measured by the radiological response rate prior to NC in patients with advanced or metastatic renal cell cancer candidates for NC.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — This study tries to clarify whether Cabozantinib could be a safe and effective preoperative treatment in patients with advanced RCC who were candidates for removing a part or all of their kidney.
  Other Names: No other intervention names

SUMMARY:
Phase II, multicenter, national, uncontrolled, multicenter, uncontrolled, phase II clinical trial for the evaluation of cabozantinib treatment prior to cytoreductive nephrectomy in patients with advanced or metastatic renal cell cancer candidates for primary tumor cytoreductive nephrectomy (NC).

DETAILED DESCRIPTION:
Metastatic Renal cell carcinoma (RCC) is a type of kidney cancer that arises in the small tubes of the kidneys and has spread to other parts of the body (advanced cancer/metastases). Patients typically have surgery to remove a part or all of their kidney (called partial or radical nephrectomy). Other treatments include chemotherapy, targeted therapy, immunotherapy and hormone therapy and may be used before or after surgery or radiotherapy.

There is no standard drug therapy given before surgery, but such preoperative therapy is used widely in the treatment of other cancer types. This approach has several potential advantages, including shrinking the tumor to help improve surgical outcomes and to help find an appropriate drug therapy.

Cabozantinib is the generic for the trade chemotherapy drug CABOMETYX™ (cabozantinib). It is known as a cancer growth inhibitor and also an angiogenesis inhibitor. Tyrosine kinases are proteins that control how cells grow and divide. By blocking the activity of these proteins in cancer cells, the medicine reduces the growth and spread of cancer.

This study tries to clarify whether Cabozantinib could be a safe and effective preoperative treatment in patients with advanced RCC who were candidates for removing a part or all of their kidney.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with locally advanced or metastatic renal cell carcinoma with a clear cell component confirmed histologically by biopsy.
2. Patients eligible for cytoreductive nephrectomy according to their surgical risk established in routine clinical practice at the site.
3. Age ≥ 18 years.
4. Patients with an ECOG (Eastern Cooperative Oncology Group) performance status of between 0 and 1.
5. Patients with appropriate organ and bone marrow function within 4 weeks prior to starting treatment with cabozantinib:

   * Leukocyte count > 4,000 cells/μL
   * Hemoglobin > 9 g/dL
   * Platelet count > 100,000/mm3
   * Serum creatinine < 2.0 mg/dL or serum creatinine clearance > 30 mL/min (according to the Cockcroft-Gault formula (Cockcroft and Gault 1976).
   * Preserved liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x upper limit of normal (ULN) in the absence of liver metastases; < 5 x ULN in the case of liver metastases.
   * Lipase < 2 x ULN. Amylase < 2 x ULN.
   * INR (international normalized ratio) and APTT (activated partial thromboplastin time) ≤ 1.5 x ULN of the site. This only applies to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation with low molecular weight heparins should maintain stable doses.
6. Patients with no radiological or clinical evidence of pancreatitis.
7. Patients with evaluable tumor disease according to the RECIST criteria 1.1 (Eisenhauer et al. 2009).
8. Patients with controlled blood pressure (systolic < 145 mmHg; diastolic blood pressure < 90 mmHg).
9. Patients who sign informed consent to participate in the study.
10. Patients may have brain metastases appropriately treated with radiation therapy and/or surgery (including radiosurgery), as long as they do not require the concomitant use of corticosteroids.

Exclusion Criteria:

1. Patients with a second active malignant tumor.
2. Patients with tumors treated in the last 2 years.
3. Pregnant or breastfeeding women.
4. Women of child-bearing potential who do not agree to use a contraceptive method during treatment. Women participating in the study should have undergone surgical sterilization, be post-menopausal, or agree to use a highly effective contraceptive method (in accordance with CTFG (clinical trial facilitation group) criteria) during the treatment period. Patients of both sexes and their partners must use effective contraception during treatment and, at least, up to four months after completing treatment. Since oral contraceptives cannot possibly be considered "effective contraceptive methods", they should be used in conjunction with another method, such as a barrier method
5. Fertile men who do not agree to use a contraceptive method during treatment. Male participants in the study should have undergone surgical sterilization, or agree to use a highly effective contraceptive method (in accordance with CTFG (clinical trial facilitation group) criteria) during the treatment period.
6. Patients with gastrointestinal disorders, including:

   * Inability to take oral medication.
   * Need for parenteral nutrition.
   * Prior surgical procedures affecting absorption.
   * Active gastrointestinal bleeding.
   * Malabsorption syndrome.
   * Gastrointestinal disorders that increase the risk of perforation.
7. Patients who have had any of the following conditions within the 12 months prior to inclusion in the study: myocardial infarction, uncontrolled angina, uncontrolled hypertension, peripheral arterial or coronary graft bypass, congestive heart failure, stroke, or transient ischemic attack.
8. Patients with tumors that invade or affect major blood vessels, gastrointestinal tract, or trachea/bronchi.
9. Patients with human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related diseases.
10. Patients with active hepatitis or hepatitis C.
11. Patients with active tuberculosis.
12. Patients with uncontrolled (Ca > 12 mg/dL) or symptomatic hypercalcemia who require continuous treatment with bisphosphonates or denosumab.
13. Patients who have undergone major surgery within 4 weeks prior to inclusion in the study.
14. Patients with active bleeding.
15. Patients with a recent episode of intestinal obstruction.
16. Patients who have previously received VEGF (vascular endothelial growth factor)-targeted therapy for advanced disease.
17. Patients who have undergone radiation therapy for bone metastases within 2 weeks prior to the first dose of cabozantinib, or any external radiation therapy within 4 weeks prior to the first dose of cabozantinib.
18. Patients who have received an allogeneic transplant or stem cells in the last 5 years.
19. Malignant tumors within 3 years before Day 1 of Cycle 1, except for those with negligible risk of metastasis or death and who have been treated with curative intent, such as cervical carcinoma in situ or localized prostate cancer treated with curative intent.
20. Patients receiving therapeutic doses of oral anticoagulants (e.g., warfarin, direct thrombin inhibitors and Factor Xa) or antiplatelet agents (e.g., clopidogrel). The use of low molecular weight heparins is allowed
21. Hypersensitivity to the active substance or to any of the excipients (exclude lactose intolerant patients since each film-coated tablet contains 46.61 mg of lactose).
22. Any other clinical condition that the physician responsible for the patient considers to be inappropriate for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Radiological response rate prior to cytoreductive nephrectomy | At 12 weeks following the start of the treatment.
  Objective response to preoperative treatment with cabozantinib, defined as the percentage of patients that reach complete or partial radiological response after a 12-week cycle of treatment with cabozantinib, defined according to the RECIST 1.1 criteria (Response Evaluation Criteria In Solid Tumors: complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD))

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo de Velasco, MD PhD, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (8):
- Spain (8):
  - Institut Català d'Oncologia. Idibell, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Valdecilla, Santander, Cantabria
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Univeristario 12 de Octubre, Madrid
  - Centro Oncológico Clara Campal - HM CIOCC, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Severo Ochoa, Madrid